CLINICAL TRIAL: NCT06371898
Title: Comparison of MORbidity of Submucosal DIssection Resection of Giant cOlon Lesions Versus Surgery: a National Multicenter Study
Brief Title: Comparison of MORbidity of Submucosal DIssection Resection of Giant cOlon Lesions Versus Surgery: a National Multicenter Study (MORDIGO)
Acronym: MORDIGO
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0088 - MORDIGO
Record Dates: First submitted 2024-04-15; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Colonic Neoplasms
Keywords: endoscopy submucosal dissection; colonic neoplasms; colonic surgery
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESD: Cohort of patients with giant colonic lesions resected by ESD, in which patients will be matched to group B
- surgery: Cohort of patients who underwent colonic surgery for T1 or T2 or in situ colon cancer

SUMMARY:
Propose a one-piece endoscopic resection such as endoscopic submucosal dissection (ESD) rather than surgery for benign lesions and superficial T1 cancers colorectal cancers offers comparable efficacy with better tolerability. This approach is all the more in the rectum, even for giant lesions lesions (over 8cm), as rectal surgery is particularly morbid, with particularly morbid, with a functional impact that can impact, whereas rectal ESD is less prone to complications fewer complications than in the colon. Colonic ESD for giant lesions is a longer and more morbid more time-consuming and morbid than for smaller lesions, the question of colonic surgery in this indication. this indication. In order to compare the morbidity data of patients of giant lesions with those of colectomy, a control group colectomy, a surgical control group will be set up, including patients including patients having undergone surgery for in situ T1 or T2 in situ colon cancer. Surgical resections of resection of benign lesions is generally not indicated not indicated and would not provide the necessary necessary for a comparison. T3 and T4 lesions with their own their own morbidity will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Group A :
* Patients from the FECCO cohort
* who have undergone ESDresection of a giant lesion, defined by a fresh specimen measuring more than 8cm long axis, of the colon
* Between September 2019 and 2022
* Major
* Patient affiliated to a social security scheme

Group B:

* Patients from the Registre des Tumeurs Digestives Registry (Brest University Hospital)
* Having undergone colectomy with lymph node dissection for intramucosal colonic adenocarcinoma, T1 or T2 colonic adenocarcinoma
* Between September 2019 and 2022
* Adults
* patient affiliated to a social security scheme

Exclusion Criteria:

* - rectal lesion ;
* patients under legal protection (guardianship, curatorship,

  ...) or deprived of liberty ;
* refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with colonic neoplasms
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-03-18 (Actual); Primary Completion 2025-06-17 (Estimated); Study Completion 2025-06-17 (Estimated)

PRIMARY OUTCOMES:
30 days severe morbidity | 30 days
  Comparison of severe morbidity (Clavien dindo ≥ IIIb) at 30 days of patients who underwent DSM for giant colonic lesion (group A) to that of patients who underwent surgery surgery equivalent to that which would be performed for such a lesion (group B)

SECONDARY OUTCOMES:
morbidity of ESD group | 30 days
comparison of morbidity in both groups | 30 days
reintervention | 30 days
stomia | 30 days
length of hospital stay | 30 days
readmission | 30 days
mortality | 30 days
risk factors for morbidity | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement